CLINICAL TRIAL: NCT01515605
Title: Molecular Biological and Moleculargenetic Monitoring of Therapy After Kidney Transplantation
Acronym: MoMoTxRes
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Tepel, Dr, Odense University Hospital
Other Study IDs: MoMoTxRes
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Transplantation Infection; Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients after kidney transplantation: Patients after kidney transplantation

SUMMARY:
Molecular monitoring is conducted in blood cells, plasma samples, urine samples and/or tissue from patients after kidney transplantation. In the present study the investigators examine the hypothesis that noninvasive diagnostic molecular monitoring can improve the outcome after transplantation.

Routine clinical and laboratory data from serum and urine are evaluated at baseline and after 0-1-2-3-4-12-16-52 weeks and 1-2-3-4-5-6-7-8-9-10 years after kidney transplantation. Mononuclear cells were obtained from the blood and transcripts of several diagnostic genes (including GATA3 (Trans-acting T-cell-specific transcription factor3), GATA4 (Trans-acting T-cell-specific transcription factor4), GAPDH (Glyceraldehyde 3-phosphate dehydrogenase), TRPC3 (Transient receptor potential cononical type3), TRPC6 (Transient receptor potential cononical type6), granzyme B, perforin, FOXP3 (Forkhead box P3), ISG15 (Interferon-stimulated gene 15), Mx1 (Interferon-induced GTP-binding protein), MMP3 (Matrix metalloproteinase-3), MMP9 (Matrix metalloproteinase-9), long-non-coding RNA, and others) are quantified using standard quantitative RT-PCR (Reverse transcription polymerase chain reaction) techniques. Proteomic analysis were performed in plasma and urine samples. Polymorphisms of selected genes are analyzed using standard techniques. Data are analyzed by descriptive statistics. Differences between groups were analyzed using Mann-Whitney test or Kruskal-Wallis-test and Dunn's multiple comparison post-test, as appropriate. Associations between variables are analyzed using regression analyses. Contingency tables are analyzed using Fisher's exact test.

DETAILED DESCRIPTION:
Molecular monitoring is conducted in blood cells, plasma samples, urine samples and/or tissue from recipients after kidney transplantation and donors. In the present study the investigators examine the hypothesis that noninvasive diagnostic molecular monitoring can improve the outcome after transplantation.

Routine clinical and laboratory data from serum and urine are evaluated at baseline and after 0-1-2-3-4-12-16-52 weeks and 1-2-3-4-5-6-7-8-9-10 years, after kidney transplantation. Mononuclear cells were obtained from the blood and transcripts of several diagnostic genes (including GATA3 (Trans-acting T-cell-specific transcription factor3), GATA4 (Trans-acting T-cell-specific transcription factor4), GAPDH (Glyceraldehyde 3-phosphate dehydrogenase), TRPC3 (Transient receptor potential cononical type3), TRPC6 (Transient receptor potential cononical type6), granzyme B, perforin, FOXP3 (Forkhead box P3), ISG15 (Interferon-stimulated gene 15), Mx1 (Interferon-induced GTP-binding protein), MMP3 (Matrix metalloproteinase-3), MMP9 (Matrix metalloproteinase-9), long-non-coding RNA, and others) are quantified using standard quantitative RT-PCR (Reverse transcription polymerase chain reaction) techniques. Proteomic analysis were performed in plasma and urine samples. Polymorphisms of selected genes are analyzed using standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients after kidney transplantation, male, female, informed consent

Exclusion Criteria:

* Deny of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplantation
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2033-03-31 (Estimated); Study Completion 2033-03-31 (Estimated)

PRIMARY OUTCOMES:
Cellular transcripts | Day1
  Transcripts and protein

SECONDARY OUTCOMES:
Cellular transcripts | Day8
  Transcripts and protein
Cellular transcripts | Day15
  Transcripts and protein
Cellular transcripts | Day22
  Transcripts and protein
Cellular transcripts | Day29
  Transcripts and protein
Plasma proteome | Day1
  Plasma Proteome
Plasma proteome | Day8
  Plasma proteome
Plasma proteome | Day15
  Plasma proteome
Plasma proteome | Day22
  Plasma proteome
Plasma proteome | Day29
  Plasma proteome
Urine proteome | Day1
  Urine proteome
Urine proteome | Day8
  Urine proteome
Urine proteome | Day15
  Urine proteome
Urine proteome | Day22
  Urine proteome
Urine proteome | Day29
  Urine proteome
Association of kidney function, glomerular filtration rate, infections, therapy | Day29
  Association of kidney function, glomerular filtration rate, infections, therapy
Association of kidney function, glomerular filtration rate, infections, therapy | Month6
  Association of kidney function, glomerular filtration rate, infections, therapy
Association of kidney function, glomerular filtration rate, infections, therapy | Month12
  Association of kidney function, glomerular filtration rate, infections, therapy

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tepel, Dr, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, DK, Denmark

IPD SHARING:
Plan to Share IPD: No